CLINICAL TRIAL: NCT02842580
Title: Randomized Phase II Study Assessing the Efficacy and Safety of 2 Therapeutic Strategies Combining Bevacizumab With Chemotherapy: De-escalation Versus Escalation in Patients With Non-pretreated Unresectable Metastatic Colorectal Cancer
Brief Title: De-escalation Chemotherapies Versus Escalation in Non Pre-treated Unresectable Patients With Metastatic Colorectal Cancer
Acronym: HIGH-LIGHT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion rythm too slow.
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 45
Record Dates: First submitted 2016-07-13; First posted 2016-07-25 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal; cancer; metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Leucovorin; Irinotecan; Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (escalation strategy - arm A) (Active Comparator): LV5FU2 (5 FLUOROURACYL)+avastin. After progression: FOLFIRI + avastin. after the 2nd progression:FOLFOX4 (eloxatine)+ avastin.
  Interventions: Drug: 5 FLUOROURACYL; Drug: acide folinique; Drug: irinotecan; Drug: Oxaliplatin; Drug: capécitabine; Drug: bevacizumab
- Experimental arm (de-escalation strategy -arm B) (Experimental): (4 cycles of FOLFOXIRI (campto) + avastin and 4 cycles of FOLFIRI + avastin) is followed by maintenance with capecitabine
  Interventions: Drug: 5 FLUOROURACYL; Drug: acide folinique; Drug: irinotecan; Drug: Oxaliplatin; Drug: capécitabine; Drug: bevacizumab

INTERVENTIONS:
Drug: 5 FLUOROURACYL — Folinic acid is administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as a 2 hr infusion.
  The 5FU bolus is administered in less than 10 minutes at 400 mg/m² (on D1). The continuous 5FU is administered IV at a dose of 2400 mg/m² over 46 hr (D1 and D2).
  The cycles will last 14 days. For this 1st line chemotherapy, the investigator has the choice of using capecitabine instead of LV5FU2; in this case the cycle lasts 21 days.
  Other Names: FLUOROURACILE EBEWE
Drug: acide folinique — 200 mg/m² if Elvorine
  Other Names: ELVORINE
Drug: irinotecan — Irinotecan is administered IV at a dose of 180 mg/m² over 90 minutes. Folinic acid is administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as an infusion over 2 hours, to be given in Y along with irinotecan.
  The 5FU bolus is administered in less than 10 minutes at 400 mg/m² (on D1). The continuous 5FU is administered IV at a dose of 2400 mg/m² over 46 hr (D1 and D2).
  The cycles will last 14 days.
  Other Names: CAMPTO
Drug: Oxaliplatin — Oxaliplatin is administered IV at a dose of 85 mg/m² over 120 minutes. Folinic acid is administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as an infusion over 2 hours, to be given in Y along with oxaliplatin.
  The 5FU bolus is administered in less than 10 minutes at 400 mg/m² (on D1). The continuous 5FU is administered IV at a dose of 2400 mg/m² over 46 hr (D1 and D2).
  The cycles will last 14 days.
  Other Names: ELOXATINE 5 mg/ml
Drug: capécitabine — For this 1st line chemotherapy, the investigator has the choice of using capecitabine instead of LV5FU2; in this case the cycle lasts 21 days.
  Other Names: XELODA
Drug: bevacizumab — Bevacizumab is administered IV at a dose of 5 mg/kg over 90 min at cycle 1, then 60 min at cycle 2 and 30 min in subsequent cycles. Bevacizumab is administered every 2 weeks before the start of chemotherapy
  Other Names: AVASTIN

SUMMARY:
The intensity of tumour response appears to be correlated with the feasibility and the duration of a therapeutic pause or of a reduced maintenance therapy maintained until progression in patients initially controlled by so-called "induction" chemotherapy. Bevacizumab combined with cytotoxic chemotherapy (5-FU, irinotecan and/or oxaliplatin) has shown that it is possible to improve the tumour response rate and patient prognosis in 1st and 2nd lines. With a very favourable safety profile , it is an excellent candidate as induction treatment and also as maintenance treatment. Prospective data from recent trials have actually demonstrated improvement in PFS and/or overall survival with bevacizumab maintenance alone or in combination with 5FU (or capecitabine) after induction chemotherapy (FOLFIRI or FOLFOX + bevacizumab).

At the same time, the maintenance of anti-angiogenic pressure after progression in 1st line metastatic has demonstrated its benefit in terms of PFS and overall survival. Bevacizumab maintenance in 2nd line metastatic, despite progression, thus appears to be a valid strategy.

DETAILED DESCRIPTION:
Thus, the objective of this work is to combine continuous blocking of angiogenesis by bevacizumab given on the first 3 metastatic lines in a randomised phase II trial evaluating a "descending" strategy of immediate optimisation by 4 cycles of FOLFOXIRI-bevacizumab and 4 cycles of FOLFIRI-bevacizumab, followed by maintenance treatment with 5FU-bevacizumab until progression (re-introduction of induction in case of progression) and evaluate an "ascending" strategy with 5FU-bevacizumab immediately followed, at progression, by the introduction of irinotecan, then oxaliplatin, with maintenance of blocking of angiogenesis by bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer, histologically proven (on primary tumour and/or metastases)
* Unresectable and non-pretreated metastases
* BRAF wild-type
* Patient considered able to receive 3 lines of chemotherapy
* At least one measurable target lesion > 1 cm according to RECIST 1.1 (Appendix 4)
* Tumour assessment according to RECIST, performed 4 weeks or less prior to randomization
* Age ≥ 18 years
* WHO performance status ≤ 2 (Appendix 5)
* No major surgery within 4 weeks prior to randomisation. Wound healing must be complete
* Life expectancy greater than 3 months
* Laboratory tests: Neutrophils ≥ 1500/mm3, platelets ≥ 100,000/mm3, haemoglobin > 9 g/dL
* Creatinine clearance > 30 mL /min (capecitabine dose modification if the creatinine clearance < 30-50 mL/min), serum creatinine < 1.25 x ULN
* Liver function tests: bilirubin < 1.25 x ULN, AST/ALT < 5 x ULN
* Women of childbearing age and men (who have sexual relations with women of childbearing age) must agree to use effective contraception without interruption throughout the duration of treatment and for 6 months after the last administration
* Signed informed consent

Exclusion Criteria:

* Patient with a potentially resectable colorectal cancer; i.e. for whom the goal of chemotherapy would be to make all metastases resectable
* Patients with symptomatic metastases
* Patient with aggressive disease and a large tumour volume
* Active gastroduodenal ulcer, wound or bone fracture
* At least one of the following laboratory values: Neutrophils <1500/mm3, platelets < 100,000/mm3, haemoglobin < 9 g/dL, total bilirubin > 1.5 N, alkaline phosphatase > 2.5 N (or > 5 N in case of hepatic involvement), serum creatinine > 1.5 N, 24 hr proteinuria > 1 g
* Chronic inflammatory bowel disease, extensive resection of the small bowel
* Clinically significant coronary artery disease or a history of myocardial infraction within the last 6 months. Uncontrolled hypertension while receiving chronic medication
* Abdominal or major extra-abdominal surgical procedure (except diagnostic biopsy) or radiation within 4 weeks before starting treatment
* Previous treatment with an anti-angiogenic or irinotecan
* Known or suspected central nervous system metastasis CNS metastases, or suspected CNS metastases
* Other previous malignancies within 5 years, except for basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix - Peritoneal macro-nodular carcinomatosis
* History of haemoptysis ≥ grade 2 (defined as ≥ 2.5 mL of bright red blood per episode) in the month prior to inclusion
* Known hypersensitivity to any component of bevacizumab or to one of the study treatments
* Active infection requiring intravenous antibiotics at start of treatment
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to treatment start
* Pregnant or breastfeeding women
* Concomitant participation in another clinical study involving a drug during the treatment phase and 30 days before starting the study treatment
* Patient unable to undergo medical treatment for geographical, social, psychological or legal reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc PHELIP, MD-PhD, Principal Investigator — CHU St Etienne
Locations (11):
- France (11):
  - Hopital Pierre Oudot - Service de Gastroenterologie, Bourgoin
  - Ch de Cholet - Service Maladies de L4Appareil Digestif Du Dr Kaasis, Cholet
  - Chd Vendee - Service D'Hge, La Roche-sur-Yon
  - Ch Annecy Genevois - Service Hge, Pringy
  - CH - Annecy Genevois, Pringy
  - Chu Robert Debre - Medecine Ambulatoire-Cancerologie, Reims
  - CHU Robert DEBRE, Reims
  - Chu Charles Nicolle - Service D'Hge, Rouen
  - Hopital Prive Saint Gregoire - Service de Radiotherapie, Saint-Grégoire
  - Chu de Saint Etienne-Hopital Nord - Service Hge, Saint-Priest-en-Jarez
  - Centre Hospitalier de St Malo - Service Hepato-Gastro-Enterologie, St-Malo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized between 15 September 2016 and 10 April 2018 by 9 french centers
Groups:
- Standard Arm (Escalation Strategy - Arm A): LV5FU2 +avastin then after progression: FOLFIRI + avastin and then after the 2nd progression:FOLFOX4 (eloxatine)+ avastin.
  5 FLUOROURACYL: administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as a 2 hr infusion.
  The 5FU bolus is administered in less than 10 minutes at 400 mg/m² (on D1). The continuous 5FU is administered IV at a dose of 2400 mg/m² over 46 hr (D1 and D2).
  Irinotecan: administered IV at a dose of 180 mg/m² over 90 minutes. Folinic acid :administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as an infusion over 2 hours, to be given in Y along with irinotecan.
  Oxaliplatin: administered IV at a dose of 85 mg/m² over 120 minutes.
  bevacizumab: administered IV at a dose of 5 mg/kg over 90 min at cycle 1, then 60 min at cycle 2 and 30 min in subsequent cycles.
  Bevacizumab is administered every 2 weeks before the start of chemotherapy
- Experimental Arm (De-escalation Strategy -Arm B): (4 cycles of FOLFOXIRI (campto) + avastin and 4 cycles of FOLFIRI + avastin) is followed by maintenance with capecitabine
  5 FLUOROURACYL: Folinic acid is administered IV at a dose of 400 mg/m² (or 200 mg/m² if Elvorine) as a 2 hr infusion.
  The 5FU bolus is administered in less than 10 minutes at 400 mg/m² (on D1). The continuous 5FU is administered IV at a dose of 2400 mg/m² over 46 hr (D1 and D2).
  acide folinique: 200 mg/m² if Elvorine
  irinotecan: administered IV at a dose of 180 mg/m² over 90 minutes.
  Oxaliplatin: administered IV at a dose of 85 mg/m² over 120 minutes.
  capécitabine: For this 1st line chemotherapy, the investigator has the choice of using capecitabine instead of LV5FU2; in this case the cycle last 21 days.
  bevacizumab: Bevacizumab is administered IV at a dose of 5 mg/kg over 90 min at cycle 1, then 60 min at cycle 2 and 30 min in subsequent cycles. Bevacizumab is administered every 2 weeks before the start of chemotherapy
Period: Overall Study
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is the ITT population meaning all the patients randomized into the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.70 (9.14) | 66.32 (10.2) | 65.99 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 11 | 10 | 21
kRAS mutation status (V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog) [Count of Participants; unit: Participants]
  Mutated | 8 | 7 | 15
  Non mutated | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective Was the Percentage of Patients Without Failure of the Strategy 16 Months After the Randomization.
Description: The failure of the strategy is defined by the following events:
  * Progression (under certain condition) using RECIST version 1.1 and defined as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed durin the study (NADIR), or a measurable increase in a nontarget lesion, or the appearance of new lesions
  * Death (all causes)
  * Toxicity leading to definitive stop of chemotherapy (oxaliplatine and/or irinotecan).
Time Frame: 16 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
Number analyzed (Participants) | 11 | 10
Participants
  No strategy failure | 7 | 4
  Strategy failure | 4 | 6

2. Secondary Outcome: Best Response Rate (Using RECIST Version 1.1)
Description: Best response derived from all the CT scans performed during treatment and based on RECIST 1.1 definition of response.
Time Frame: At 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
Number analyzed (Participants) | 11 | 10
Participants
  Complete response | 0 | 1
  Partial response | 3 | 6
  Stability | 7 | 2
  Progression | 0 | 1
  Non evaluable | 1 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of the patient's inclusion to the patient's death (all causes). For alive patients the date of the latest news was taken into account
Time Frame: Up to 3 years after the treatment start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
Number analyzed (Participants) | 11 | 10
months | 31.08 [15.51 to NA] — Upper limit of the confidence interval was not reached at the time of the study analysis because less than 75% of the patients died at the time of the analysis | 33.80 [3.68 to NA] — Upper limit of the confidence interval was not reached at the time of the study analysis because less than 75% of the patients died at the time of the analysis

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The progression-free survival is the time from inclusion to the first radiological progression or death (all causes). For patients alive without progression date of last news will be considered.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed durin the study (NADIR), or a measurable increase in a nontarget lesion, or the appearance of new lesions
Time Frame: up to 24 months after randomization
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
Number analyzed (Participants) | 11 | 10
months | 8.24 [4.27 to 12.19] | 13.22 [2.27 to 23.49]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment for each patient. The mean time of treatment was 16 months. After patient could have another treatment and patients were followed only for overall survival up to 3 years after the treatment start.
Arm/Group | Standard Arm (Escalation Strategy - Arm A) | Experimental Arm (De-escalation Strategy -Arm B)
All-Cause Mortality (participants affected / at risk) | 6/11 | 5/10
Serious Adverse Events (participants affected / at risk) | 4/11 | 0/10
Other Adverse Events (participants affected / at risk) | 10/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Arm (Escalation Strategy - Arm A) (N=11) | Experimental Arm (De-escalation Strategy -Arm B) (N=10)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Arm (Escalation Strategy - Arm A) (N=11) | Experimental Arm (De-escalation Strategy -Arm B) (N=10)
Hypertension (Cardiac disorders) | 2 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 5
Proteinuria (Renal and urinary disorders) | 4 | 4
Cephalgia (Nervous system disorders) | 2 | 2
Sensitive peripheral neuropathy (Nervous system disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Mucositis (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 9 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Thromboembolic event (Vascular disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 5 | 2
Anemia (Investigations) | 7 | 8
Total Bilirubin increased (Investigations) | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 9 | 6
White blood cell count decreased (Investigations) | 3 | 3
Neutrophils decreased (Investigations) | 5 | 0
Phosphatases Alcalines increased (Investigations) | 8 | 6
Thombopenia (Investigations) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkaliemia (Metabolism and nutrition disorders) | 5 | 3
Hypoalbuminumia (Metabolism and nutrition disorders) | 3 | 0
Asthenia (General disorders) | 8 | 8
Fever (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT02842580/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02842580/SAP_001.pdf